CLINICAL TRIAL: NCT07095244
Title: Pediatric Outcomes and Recovery With Peri-Operative Iron Supplement Evaluation (PORPOISE)
Brief Title: Pediatric Outcomes and Recovery With Peri-Operative Iron Supplement Evaluation
Acronym: PORPOISE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: BC Children's Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Teresa Skelton, Clinical Associate Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H25-00010
Record Dates: First submitted 2025-05-26; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Varus-Derotation Osteotomy Surgery; Iron-deficiency Anemia; Pelvic Osteotomy Surgery; Cerebral Palsy
Keywords: Varus-derotation osteotomy; Anemia; Iron deficiency; Nutrition; Perioperative blood management
MeSH Terms: conditions — Anemia, Iron-Deficiency; Cerebral Palsy; Anemia; Iron Deficiencies | interventions — Iron-Dextran Complex

STUDY DESIGN:
Intervention Model Description: All participants who are enrolled prospectively will receive comprehensive nutrition management, which includes a blood test. Participants will have their blood work done prior to initiating nutrition intervention for iron-deficiency (two tubes containing 1 to 2 ml each). If patients are determined to be iron-deficient or anemic, they will be prescribed iron supplementation. All patients will receive comprehensive nutrition management from a clinical dietician during the months leading up to their procedure (up to 12 months preoperatively). Patients will have their blood re-tested in the operating room before surgery (after the induction of anesthesia).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Prospective (Iron Supplementation) (Experimental): Patients scheduled for VDRO and/or pelvic osteotomy surgery who are aged 0 to 18 years old (n = 50-60). Note that the investigators will include patients who do or do not have a diagnosis of a neuromotor condition. All patients will be evaluated by the dietitian and have screening lab work to evaluate for iron deficiency at initial consultation. If lab results show that iron supplementation is required, patients will be allocated to the iron supplementation arm and will receive a prescription for iron supplementation, education on non-pharmacological methods to enhance iron intake and comprehensive nutrition management.
  Interventions: Dietary Supplement: Iron Supplement; Dietary Supplement: Comprehensive Nutrition Management
- Historical (No Intervention): All patients who had VDRO and/or pelvic osteotomy surgery between February 2022 and December 2024 who are aged 0 to 18 years old (n = 100-120). These participants will be enrolled as comparators and receive no intervention, as their surgery has passed.
- Prospective (No Iron Supplementation) (Experimental): Patients scheduled for VDRO and/or pelvic osteotomy surgery who are aged 0 to 18 years old (n = 50-60). Note that the investigators will include patients who do or do not have a diagnosis of a neuromotor condition. All patients will be evaluated by the dietitian and have screening lab work to evaluate for iron deficiency at initial consultation. If lab results show adequate iron levels, patients will be allocated to the "no iron supplementation" arm and will only receive comprehensive nutrition management, without an iron supplementation prescription.
  Interventions: Dietary Supplement: Comprehensive Nutrition Management

INTERVENTIONS:
Dietary Supplement: Iron Supplement — FeraMAX Pd powder 15: NPN 80109337 FeraMAX Pd Therapeutic 150 capsules: NPN 80075623 (for an adolescent that can swallow capsules)
  Arms: Prospective (Iron Supplementation)
Dietary Supplement: Comprehensive Nutrition Management — Standard nutrition care will depend on the results of the nutrition assessment, as well as underlying conditions, and will be performed regardless of iron supplementation. The intervention will be at the discretion of the dietician but may include; diet education, recommendations for vitamin and mineral supplements, optimization of tube feeds (if the child is tube fed), high protein or high energy diet education if the child is underweight, dddition of oral nutrition supplements (i.e., Pediasure or Ensure) to promote weight gain in orally fed children, discussion surrounding enteral feeding (for children who are orally fed, but severely malnourished and cannot meet their nutritional needs by mouth).
  Other Names: Standard Nutrition Care
  Arms: Prospective (Iron Supplementation); Prospective (No Iron Supplementation)

SUMMARY:
Varus-derotation osteotomy (VDRO) is a surgery to prevent or address hip displacement in children. Many children having this surgery have cerebral palsy or other neuromotor disorders, who have a higher rate of malnutrition, including low iron or anemia. This can affect their surgical outcomes, such as increasing their need for blood transfusions. This project aims to develop a preoperative nutritional program for VDRO patients, to improve their surgical outcomes and decrease their need for transfusions. This may include taking iron supplementation for patient with low iron or anemia. Participants will undergo a nutrition program before their surgery.

DETAILED DESCRIPTION:
Purpose:

The investigators aim to establish a multidisciplinary pathway for all patients scheduled for varus-derotation osteotomy (VDRO) surgery that incorporates comprehensive nutrition management and iron deficiency anemia assessment and management. The goal is to determine whether patients with nutritional optimization will experience improved care, including a decreased risk of adverse outcomes and improved surgical outcomes.

Hypothesis:

The primary hypothesis is that a comprehensive nutritional prehabilitation intervention for iron deficiency anemia before pediatric varus-derotational osteotomy (VDRO) surgery will decrease the risk blood transfusion, as shown by a lower incidence of blood transfusions, during the preoperative period. The investigators also aim to show that this program will improve other perioperative surgical outcomes and will be feasible and acceptable to families.

Justification:

VDRO, a surgical procedure designed to prevent or address hip displacement, is a lengthy procedure (>4 hours), with risk of blood transfusion from 10-25%. VDRO patients often present with complex medical conditions and require multidisciplinary care. Malnutrition contributes to morbidity but is rarely highlighted by the perioperative team. Similarly, while patient blood management programs are standard perioperative care for adults, their implementation in pediatrics is limited. Estimates of iron-deficiency anemia in Canadian children range from 12-64%, without considering medically complex patients at high risk of malnutrition. Preoperative anemia raises the risk of in-hospital mortality for pediatric surgical patients. BC Children's Hospital treats 30-35 VDRO patients annually. The investigators aim to establish a multidisciplinary nutritional and prehabilitation program for elective VDRO patients (with and without neuromotor conditions) that includes comprehensive nutrition and iron deficiency anemia management.

Objectives:

(1) Study the integration of blood management into the nutritional care of patients having VDRO surgery and determine whether it improves perioperative outcomes; (2) evaluate the program's operational feasibility and its acceptability among patients' families; (3) apply the findings to other elective surgical interventions, such as neuromuscular scoliosis surgery.

Research Design:

The investigators will conduct a prospective observational study to evaluate this comprehensive nutritional prehabilitation program over a 24-month period and compare outcomes against a historical cohort from February 2022 to December 2024 using propensity score matching. The primary outcome will be the percentage of patients transfused during the perioperative stay. Secondary perioperative outcomes will include anemia, iron levels, length of hospital stay, and surgical complications such as pressure sores. The investigators will recruit all patients 0-18 years scheduled to undergo VDRO and/or pelvic osteotomy, unless they have undergone a surgical intervention or received a nutritional intervention that includes iron within the previous 3 months. All patients will be evaluated by the dietitian and have screening lab work to evaluate for iron deficiency at initial consultation. If required, patients will receive a prescription for iron supplementation and education on non-pharmacological methods to enhance iron intake. Longitudinal online surveys will assess compliance/tolerance and family satisfaction with the program. Further feedback will be obtained in optional semi-structured interviews.

Iron Supplementation Intevntion:

Feramax (or other iron polysaccharide complex) will be prescribed as it is most used in practice due to its fewer gastrointestinal side effects, ability to be taken with food, and lack of requirement for stomach acid for absorption, making it suitable for patients receiving gastrojejunostomy feedings. The typical dose of iron for pediatric patients with deficiency is 3-6 mg/kg, up to a maximum of 150 mg/day. Other possible nutritional interventions may include recommending supplements (most commonly calcium/Vitamin D and occasionally a multivitamin), optimizing tube feeds, and providing dietary education.

Standard Nutrition Intervention:

Standard nutrition care will depend on the results of the nutrition assessment, as well as underlying conditions, and will be performed regardless of iron supplementation. The intervention will be at the discretion of the dietician but may include components of the following non-exhaustive list.

1. Diet education regarding general healthy diet and nutrition for bone health (for generally healthy orally fed patients).
2. Recommendations for vitamin and mineral supplements as needed (based on estimated intake from diet or tube feeds. This may include a multivitamin, calcium and/or Vitamin D.
3. Optimization of tube feeds (if the child is tube fed).
4. High protein or high energy diet education if the child is underweight, but capable of achieving their nutritional needs by increasing oral intake.
5. Addition of oral nutrition supplements (i.e., Pediasure or Ensure) to promote weight gain in orally fed children.
6. Discussion surrounding enteral feeding (for children who are orally fed, but severely malnourished and cannot meet their nutritional needs by mouth). The orthopedic surgeon may refer the patient to general surgery, or the family may ask their pediatrician for a referral.

Statistical Analysis The investigators will recruit a convenience sample of participants over a two-year period (n~50); the investigators will propensity-score match each prospective participant to two historical controls based on age, sex, gross motor function classification system score, ASA physical status score, and procedure booking code. Transfusion rates between the baseline period and the intervention period will be compared using Fisher's exact test. Semi-structured interviews will be analyzed using a grounded theory-based qualitative approach.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for VDRO and/or pelvic osteotomy surgery (prospective cohort)
* All patients who had VDRO and/or pelvic osteotomy surgery between February 2022 and December 2024 (historical cohort)
* Ages 0-18 years old

Note that the investigators will include patients who do or do not have a diagnosis of a neuromotor condition. The investigators may not include patients who are enrolled in other conflicting research studies.

Exclusion Criteria:

* Patients who have undergone a major surgical intervention in the last 3 months
* Patients who have received a nutritional intervention that includes iron testing and treatment within the last 3 months
* Patients in whom oral/enteral iron supplementation is contraindicated
* Patients who have a bleeding disorder
* Patients taking erythropoietin
* Patients who cannot read and understand English*

  * Patients and their families who cannot read and understand English will be excluded from the study because the surveys and interviews are conducted in English. These patients will still have access to the same nutrition management and interventions as study participants.

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Decreased incidence of blood transfusion | From surgery start time to discharge from hospital.
  A comprehensive nutritional prehabilitation intervention for iron deficiency anemia before pediatric VDRO surgery will decrease the risk of requiring a blood transfusion, as shown by a decreased incidence of blood transfusions, in the perioperative period.

SECONDARY OUTCOMES:
Resolution of anemia | From baseline to 12 months post-op.
  As per the Government of British Columbia guidelines, the investigators will consider iron supplementation for blood Ferritin < 20 mcg/L for participants aged 0 to 2 years old and < 30 mcg/L for participants aged 3 years or older. Cases where Ferritin is < 100 mcg/L, but Transferrin saturation is <20% will also be considered for iron supplementation.
  Participants who fall into the above categories at the time of their initial nutrition consultation, but no longer do at the time of surgery, will have their anemia considered "resolved".
Increased Iron Levels | From baseline to 12 months post-op.
  Iron supplementation (if prescribed/necessary) will increase iron levels as proven by a comparison between the blood test at the time of the nutrition consultation and the time of surgery, as shown by Ferritin levels.
Lower incidence of surgical site infection and pressure wounds | From the day of surgery to 30 days post-op.
  The investigators will compare the number and type of adverse outcomes (including surgical site infection and pressure wounds) between the retrospective (no intervention) and prospective (iron supplementation and/or nutrition management) groups.
Decreased hospital length of stay | From the date of surgery until the date of hospital discharge.
  Acute inpatient length of stay (days) between retrospective (no intervention) and prospective (iron supplementation and/or nutrition management) groups.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Skelton, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data for concern that patients may be identified.

REFERENCES:
- [Background] Luo J, West NC, Pang S, Robillard JM, Page P, Chadha NK, Gan H, Correll LR, Ridgway R, Broemling N, Gorges M; Pediatric Pain Prediction Collaboration. Parental Perspectives on Pediatric Surgical Recovery: Narrative Analysis of Free-Text Comments From a Postoperative Survey. JMIR Perioper Med. 2024 Dec 20;7:e65198. doi: 10.2196/65198. PMID 39705676
- [Background] Lin Y. Preoperative anemia-screening clinics. Hematology Am Soc Hematol Educ Program. 2019 Dec 6;2019(1):570-576. doi: 10.1182/hematology.2019000061. PMID 31808909
- [Background] Tan GM, Murto K, Downey LA, Wilder MS, Goobie SM. Error traps in Pediatric Patient Blood Management in the Perioperative Period. Paediatr Anaesth. 2023 Aug;33(8):609-619. doi: 10.1111/pan.14683. Epub 2023 May 5. PMID 37144721
- [Background] Faraoni D, DiNardo JA, Goobie SM. Relationship Between Preoperative Anemia and In-Hospital Mortality in Children Undergoing Noncardiac Surgery. Anesth Analg. 2016 Dec;123(6):1582-1587. doi: 10.1213/ANE.0000000000001499. PMID 27870741
- [Background] Hartfield D. Iron deficiency is a public health problem in Canadian infants and children. Paediatr Child Health. 2010 Jul;15(6):347-50. doi: 10.1093/pch/15.6.347. No abstract available. PMID 21731416
- [Background] Goobie SM, Faraoni D. Perioperative paediatric patient blood management: a narrative review. Br J Anaesth. 2025 Jan;134(1):168-179. doi: 10.1016/j.bja.2024.08.034. Epub 2024 Oct 24. PMID 39455307
- [Background] Goel R, Cushing MM, Tobian AA. Pediatric Patient Blood Management Programs: Not Just Transfusing Little Adults. Transfus Med Rev. 2016 Oct;30(4):235-41. doi: 10.1016/j.tmrv.2016.07.004. Epub 2016 Aug 1. PMID 27559005
- [Background] DiFazio RL, Glader LJ, Tombeno R, Lawler K, Friel K, Brustowicz RM, Shore BJ. Team Approach: The Perioperative Management of Reconstructive Hip Surgery for the Non-Ambulatory Child with Cerebral Palsy and Spastic Hip Disease. JBJS Rev. 2020 Jul;8(7):e1900185. doi: 10.2106/JBJS.RVW.19.00185. PMID 32678539
- [Background] Butler LR, Dominy CL, White CA, Mengsteab P, Lin E, Allen AK, Ranade SC. Risk factors for 90-day readmission and prolonged length of stay after hip surgery in children with cerebral palsy. J Orthop. 2023 Mar 2;38:14-19. doi: 10.1016/j.jor.2023.03.002. eCollection 2023 Apr. PMID 36925762
- [Background] Fontanals M, O'Leary JD, Zaarour C, Skelton T, Faraoni D. Preoperative anemia increases the risk of red blood cell transfusion and prolonged hospital length of stay in children undergoing spine arthrodesis surgery. Transfusion. 2019 Feb;59(2):492-499. doi: 10.1111/trf.15055. Epub 2018 Nov 30. PMID 30499592
- [Background] Papadopoulos A, Ntaios G, Kaiafa G, Girtovitis F, Saouli Z, Kontoninas Z, Diamantidis MD, Savopoulos C, Hatzitolios A. Increased incidence of iron deficiency anemia secondary to inadequate iron intake in institutionalized, young patients with cerebral palsy. Int J Hematol. 2008 Dec;88(5):495-497. doi: 10.1007/s12185-008-0191-3. Epub 2008 Nov 11. PMID 18991057
- [Background] Le Roy C, Barja S, Sepulveda C, Guzman ML, Olivarez M, Figueroa MJ, Alvarez M. Vitamin D and iron deficiencies in children and adolescents with cerebral palsy. Neurologia (Engl Ed). 2021 Mar;36(2):112-118. doi: 10.1016/j.nrl.2017.11.005. Epub 2018 Jan 17. English, Spanish. PMID 29342407
- [Background] Jevsevar DS, Karlin LI. The relationship between preoperative nutritional status and complications after an operation for scoliosis in patients who have cerebral palsy. J Bone Joint Surg Am. 1993 Jun;75(6):880-4. doi: 10.2106/00004623-199306000-00008. PMID 8314827
- [Background] Ruzbarsky JJ, Beck NA, Baldwin KD, Sankar WN, Flynn JM, Spiegel DA. Risk factors and complications in hip reconstruction for nonambulatory patients with cerebral palsy. J Child Orthop. 2013 Dec;7(6):487-500. doi: 10.1007/s11832-013-0536-1. Epub 2013 Oct 15. PMID 24432112
- [Background] Nazareth A, Shymon SJ, Andras L, Goldstein RY, Kay RM. Impact of tranexamic acid use on blood loss and transfusion rates following femoral varus derotational osteotomy in children with cerebral palsy. J Child Orthop. 2019 Apr 1;13(2):190-195. doi: 10.1302/1863-2548.13.180143. PMID 30996744
- [Background] Compton E, Goldstein RY, Nazareth A, Shymon SJ, Andras L, Kay RM. Tranexamic acid use decreases transfusion rate in children with cerebral palsy undergoing proximal femoral varus derotational osteotomy. Medicine (Baltimore). 2022 Jan 14;101(2):e28506. doi: 10.1097/MD.0000000000028506. PMID 35029205
- [Background] Bouwhuis CB, van der Heijden-Maessen HC, Boldingh EJ, Bos CF, Lankhorst GJ. Effectiveness of preventive and corrective surgical intervention on hip disorders in severe cerebral palsy: a systematic review. Disabil Rehabil. 2015;37(2):97-105. doi: 10.3109/09638288.2014.908961. Epub 2014 Apr 14. PMID 24731007

DOCUMENTS (4):
  • Study Protocol and Statistical Analysis Plan (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT07095244/Prot_SAP_000.pdf
  • Informed Consent Form: Family Consent Form (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT07095244/ICF_001.pdf
  • Informed Consent Form: Child Assent Form (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/44/NCT07095244/ICF_002.pdf
  • Informed Consent Form: Adolescent Assent Form (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT07095244/ICF_003.pdf